CLINICAL TRIAL: NCT04989829
Title: A Single-centre, One-arm, Open-label, Fixed-sequence Study to Evaluate the Effect of Omeprazole on the Pharmacokinetics of SHR6390 in Healthy Male and Female Subjects
Brief Title: Effect of Omeprazole on the Pharmacokinetics of SHR6390 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: SHR6390-I-113
Record Dates: First submitted 2021-08-03; First posted 2021-08-04 (Actual); Last update posted 2023-06-08 (Actual); Status verified 2023-06

CONDITIONS: Advanced Solid Tumor

STUDY DESIGN:
Intervention Model Description: The study is a single-center, open, single-dose, Fixed-sequence clinical trial.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment group (Experimental)
  Interventions: Drug: SHR6390、Omeprazole

INTERVENTIONS:
Drug: SHR6390、Omeprazole — SHR6390 tablet single dose、Omeprazol single dose.

SUMMARY:
This is a one-arm, fixed-sequence study to compare the pharmacokinetic profiles of SHR6390 in absence and presence of prior administration of proton pump inhibitor Omeprazole. The increased gastric pH achieved by the treatment with multiple doses of Omeprazole might affect the absorption process of SHR6390.

ELIGIBILITY:
Inclusion Criteria:

1. Sign the informed consent before the trial, and fully understand the trial content, process and possible adverse reactions;
2. Ability to complete the study as required by the protocol;
3. Healthy male or female subjects aged 18 to 45 (including 18 and 45) at the date of signing the informed consent;
4. Subjects shall ake effective contraceptive measures voluntarily within 7 months from the date of signing the informed consent form to the date of the last medication. Serum HCG test of fertile women before the study must be negative;
5. Male body weight ≥ 50 kg, female body weight ≥ 45 kg, and body mass index (BMI) within the range of 19 ~ 26 kg /m2 (including 19 and 26);
6. Healthy subjects identified by a detailed medical history;
7. Full physical examinations, including blood pressure and pulse rate measurement, 12-lead ECG or clinical laboratory test, are normal or abnormal but have no clinical significance.

Exclusion Criteria:

1. Blood donation or loss≥400 mL within 3 months prior to screening, or blood donation or loss≥200 mL, or blood transfusion within 1 months before screening;
2. Participating in any clinical trial or taking drugs that might damage organs within 3 months before screening;
3. Surgeries in the previous 6 months before screening;
4. Use of vaccines or biologicals within 2 weeks prior to screening;
5. Allergic constitution;
6. History of drug abuse or alcoholism, or positive for nicotine, alcohol and drug tests;
7. History of myocarditis, coronary heart disease, arrhythmia, stroke and so on, or 12 lead ECG demonstrating a corrected QT by Fridericia (QTcF) interval ≥450 msec;
8. With dysphagia or history of gut disease or surgery (gastrectomy, enterectomy, sleeve gastrectomy, etc) possibly affecting drug absorption;
9. Uncontrolled gut disease, such as peptic ulcer, colitis, pancreatitis, etc;
10. History of chronic kidney disease, renal insufficiency, anemia of renal failure, or creatinine clearance rate (CLCr) < 80 mL/min, or serum creatinine ≥ ULN.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2021-12-27 (Actual); Primary Completion 2022-01-26 (Actual); Study Completion 2022-02-14 (Actual)

PRIMARY OUTCOMES:
Cmax | from Day1 to Day7after the first dose and from Day17 to Day23 after the second dose
  Maximum observed serum concentration (Cmax) for SHR6390 after Single dose.
AUC0-t | from Day1 to Day7after the first dose and from Day17 to Day23 after the second dose
  Area under the plasma concentration versus time curve (AUC0-t) for SHR6390 after Single dose
AUC0-∞ | from Day1 to Day7after the first dose and from Day17 to Day23 after the second dose
  Area under the plasma concentration versus time curve (AUC0-∞) for SHR6390 after Single dose

SECONDARY OUTCOMES:
Tmax | from Day1 to Day7after the first dose and from Day17 to Day23 after the second dose
  Time to maximum observed serum concentration (Tmax) for SHR6390 after Single dose
T1/2 | from Day1 to Day7after the first dose and from Day17 to Day23 after the second dose
  Time to elimination half-life (T1/2) for SHR6390 after Single dose.[Time Frame
CL/F | from Day1 to Day7after the first dose and from Day17 to Day23 after the second dose
  Apparent oral clearance (CL/F) for SHR6390 after Single dose
Vz/F | from Day1 to Day7after the first dose and from Day17 to Day23 after the second dose
  Apparent Volume of Distribution (Vz/F) SHR6390 after Single dose
Number of subjects with adverse events and severity of adverse events | from Day1 to Day30 after the first dose

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Xuhui Central Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided